CLINICAL TRIAL: NCT01445444
Title: Habit Reversal Training for Children and Adolescents With Trichotillomania: A Controlled Trial
Brief Title: Habit Reversal Training for Children and Adolescents With Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Adam Lewin, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRT/TTM
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Trichotillomania
Keywords: Habit Reversal Training; Hair Pulling; Children; Trich; cognitive behavioral therapy; TTM; psychotherapy
MeSH Terms: conditions — Trichotillomania; Trichomonas Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HRT group (Experimental): This group receives habit reversal training immediately.
  Interventions: Behavioral: Habit Reversal Training
- TAU group (Active Comparator): This group receives treatment as usual for 8 weeks.
  Interventions: Behavioral: Habit Reversal Training

INTERVENTIONS:
Behavioral: Habit Reversal Training — * 8 weekly therapy sessions lasting 50 minutes based on the protocol outlined by Woods (2001).
  * The overall focus of treatment is to provide patients with tools to help them manage and reduce hair-pulling.
  * components:
  * Session 1. (a) to develop an understanding of the subject's hair-pulling through an initial interview; and (b) to establish a protocol for ongoing assessment.
  * Session 2. implement habit reversal, including awareness training, competing response training, and social support.
  * Sessions 3-8. For subjects with a single hair-pulling site, Session 3 will review and practice HRT procedures and name solutions to problems that may have arisen. For those with multiple hair-pulling sites, treatment will be reviewed for the first site in the hierarchy.
  Other Names: Trichotillomania; Hair pulling; TTM

SUMMARY:
The purpose of the current study is:

1. To evaluate the effectiveness of a habit reversal training (HRT) approach for children ages 7 to 17 years of age inclusive with a diagnosis of trichotillomania.
2. To explore factors that may relate to symptom severity, treatment outcome, and psychosocial impairment (e.g., specific symptom presence, co-morbidity, emotional regulation).

DETAILED DESCRIPTION:
The purpose of this research study is to further investigate how well Habit Reversal Training (HRT) works to reduce hair-pulling symptoms in children and adolescents with trichotillomania (TTM).

All children will have the option to receive 8 weekly HRT sessions. Half of all children will be chosen at random to receive these sessions immediately following the pre-assessment and the remaining half will receive them after eight weeks (TAU condition). These sessions will focus developing skills for managing TTM and to decrease hair pulling. Such skills may include teaching your child to replace hair-pulling with another behavior. In the TAU condition, participants will seek the treatment in the community, with the option of receiving HRT treatment sessions at the end of the study.

Participants in both groups will undergo four assessments in total (1) Pre-Assessment; (2) Post-treatment Assessment; (3) One-month Follow-up; (4)Three-month Follow-up. These assessments will involve several interviews that ask about different psychological symptoms that your child experiences such as sadness, anxiety, and TTM.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient children between the ages of 7-17 years.
* Meets DSM-IV criteria for a primary diagnosis of TTM
* English speaking

Exclusion Criteria:

* Lifetime DSM-IV bipolar, schizophrenia, or schizoaffective disorder, or substance abuse in past 6 months.
* A diagnosis of an autism spectrum disorders, mental retardation, or conduct disorder
* 1) Current clinically significant suicidal intent, or 2) individuals who have engaged in suicidal behaviors within 6 months
* Receiving concurrent psychotherapy or behavioral interventions. Families will have the option of discontinuing such services to enroll in the study. Those randomized to treatment as usual (TAU) will be able to continue or initiate psychosocial interventions whereas those randomized to HRT will not receive other interventions concurrent with HRT.
* Any change in established psychotropic medication (e.g., antidepressants, anxioloytics) within 4 weeks before study enrollment, any change in antipsychotics within 3 weeks prior to the screening assessment, any change in fluoxetine or atamoxetine within 6 weeks of study enrollment, and any change in alpha-2 agonists or stimulants within 1 week of study enrollment. Those randomized to TAU may make medication changes following randomization, including starting a medication; those randomized to HRT will remain stable on medications during the study.
* Unwillingness of parents to make the commitment to accompany their child for multiple study visits, unwillingness to take part in randomization, inability to attend weekly sessions as therapist availability allows, inability to attend assessment visits.
* Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Massachusetts General Hospital Hairpulling Scale (MGHHS) | 5 months
  This measure assesses the number of hair-pulling urges, the intensity of the urges, the ability of the patients to distract themselves from the urge to pull their hair, the number of hair-pulling incidents, attempts to resist hair-pulling, the ability to resist hair-pulling, and feeling uncomfortable about hair-pulling. Individual items are rated for severity from 0 (no symptoms) to 4 (extreme symptoms).

SECONDARY OUTCOMES:
NIMH-TIS | 5 months
  The NIMH-TIS is a clinician rated scale (0-10 rating) measuring overall impairment produced by the time spent pulling or concealing damage, ability to control pulling, severity of alopecia, interference, and incapacitation caused by the pulling.

CONTACTS AND LOCATIONS:
Overall Officials: Adam B Lewin, Ph.D., Principal Investigator — University of South Florida; Omar Rahman, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- Rothman Center for Pediatric Neuropsychiatry, St. Petersburg, Florida, United States